CLINICAL TRIAL: NCT04664985
Title: Evaluation of Mucogyne® Ovule in Vulvovaginal Dryness Management in Women Treated by Brachytherapy and/or Radiotherapy for Endometrial or Cervical Cancer.
Acronym: HYDRAMUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratoires IPRAD (Industry)
Collaborators: Créapharm (Unknown); Institut Alfred Fournier (Unknown); Axonal-Biostatem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPR_HYDRAMUC_17
Record Dates: First submitted 2020-11-18; First posted 2020-12-11 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Vaginal Disease
Keywords: vaginal dryness
MeSH Terms: conditions — Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: 80 women with endometrial cancer or Cervical cancer will be recruited over 8 months, 40 being randomized in the Mucogyne® arm, the 40 others in the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mucogyne® (Active Comparator): The dosage during the study will be 1 Mucogyne® ovule per day at bedtime for 10 days and then 1 ovule every 2 days until the end of the 3-month follow-up.
  Interventions: Device: Mucogyne® ovule
- Control (No Intervention): No treatment for this arm.

INTERVENTIONS:
Device: Mucogyne® ovule — hyaluronic acid, vaginal ovule
  Arms: Mucogyne®

SUMMARY:
Randomized, open-label, national (France), multicenter, prospective clinical study, to evaluate the superiority of Mucogyne® ovules over the control group on vaginal health (including hydration) in women treated by brachytherapy and/or radiotherapy for endometrial or cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18
* hysterectomized patient with endometrial cancer (stage I, stage II and histological type I, without chemotherapy, with brachytherapy and/or radiotherapy) OR patient with cervical cancer (stage IA2 and IB1 with emboli or positive lymphadenopathy and IB2 stages with or without chemotherapy, with brachytherapy and / or radiotherapy)
* Only for patients with cervical cancer, premenopausal and non-hysterectomized: patient on contraception at least one month before V0 and throughout the study
* Only for patients with cervical cancer: complete remission
* Patient capable of receiving and understanding information related to the study, giving informed written consent, and easily completing a quality of life questionnaire
* Patient affiliated to the French social security system

Exclusion Criteria:

* Patient with clinically observed vulvovaginal infections
* Patient with endometrial cancer treated with chemotherapy
* Patient already participating in another study
* Patient under legal protection, or under guardianship or curatorship
* Only for patients with cervical cancer: local treatment with estrogen
* Only for patients with cervical cancer, premenopausal and non-hysterectomized: pregnancy (pregnancy test to be performed at V0)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal Health Index (VHI) change from inclusion to end of study | 3 Months
  Each parameter is evaluated from 1 (worst) to 5 (best/normal):
  * vaginal elasticity,
  * vaginal secretion volume,
  * vaginal pH,
  * epithelial mucous membrane integrity,
  * vaginal hydration/lubrication.
  The sum of points for each parameter gives the VHI, from 5 (worst) to 25 (best/normal)

SECONDARY OUTCOMES:
Vaginal mucosa scarring evolution | 3 Months
  Evolution of scarring of the vaginal mucosa by a composite score:
  * visualization of the hysterectomy scar (not visible / visible) for endometrial cancer patients OR visualization of the cervix (not visible / visible) for cervical cancer patients,
  * presence or absence of vaginal adhesions / cohalescences (walls and bottom of the vagina ),
  * collapse of adhesions to touch (Y / N),
  * edema / redness of vaginal mucosa (indicative of inflammation),
  * pain caused by pressure (Y / N),
  * bleeding caused by contact (none / moderate / severe)
Time to additional local treatment administration | 3 Months
Patient Global Impression of Change (PGIC) on vaginal health | 3 Months
  Auto-evaluation: score from 1 (very much improved) to 7 (very much worse) on vaginal health related to the study intervention
Symptoms (pain, dyspareunia, vaginal pruritis, vulvovaginal dryness) evolution | 3 Months
  Auto-evaluation of the symptoms: pain, dyspareunia, vaginal pruritis, vulvovaginal dryness on Visual Analogic Scale (VAS) of 10mm
  Patient indicates where she locates the intensity of the symptom from 0mm (no symptom) to 10mm (worst intensity)
VHI change at each visit | 3 Months
  Each parameter is evaluated from 1 (worst) to 5 (best/normal):
  * vaginal elasticity,
  * vaginal secretion volume,
  * vaginal pH,
  * epithelial mucous membrane integrity,
  * vaginal hydration/lubrication. The sum of points for each parameters gives the VHI, from 5 (worst) to 25 (best/normal)
Vaginal flora composition (Nugent score) evolution | 3 Months
  Measured on vaginal sample collected at inclusion, 1 month and 3 months
Complications and adverse events | 3 Months
  Complications and adverse events related to study intervention
Patient satisfaction questionnaire at the end of study | 3 Months
  All patients (both arms) will be asked about their satisfaction on the treatment of their vulvogainal symptoms during the study will be assessed using a 5-point Likert scale :
  "At the end of this study, how would you rate your level of satisfaction with the treatment of your vulvovaginal symptoms? Very satisfactory / Satisfactory / Moderate / Poor / Very Poor"

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Chru Besancon - Site 002, Besançon
  - Leon Berard - Site 007, Lyon
  - Institut de Cancerologie de Lorraine - Site 004, Nancy
  - Chu Nantes - Site 003, Nantes
  - Chu Caremeau - Site 001, Nîmes
  - Clinique Pasteur - Site 005, Toulouse
  - Institut Gustave Roussy - Site 006, Villejuif